CLINICAL TRIAL: NCT00143611
Title: A Pivotal, Multicenter, Multinational, Randomized, Double-Blind, Placebo-Controlled Study To Evaluate The Efficacy And Safety of TAK-242 in Adults With Severe Sepsis
Brief Title: Efficacy & Safety of Resatorvid in Adults With Severe Sepsis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-04-TL-242-011; 2005-003561-16 (EudraCT Number); U1111-1127-5919 (Registry Identifier: WHO); DOH-27-0406-1213 (Registry Identifier: SANCTR)
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Sepsis
Keywords: Shock, Septic; Sepsis Syndrome; Respiratory Insufficiency; SIRS (Systemic Inflammatory Response Syndrome); Respiratory Failure; Drug Therapy
MeSH Terms: conditions — Sepsis; Shock, Septic; Systemic Inflammatory Response Syndrome; Respiratory Insufficiency | interventions — ethyl 6-(N-(2-chloro-4-fluorophenyl)sulfamoyl)cyclohex-1-ene-1-carboxylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Resatorvid 1.2 mg/kg/day (Experimental)
  Interventions: Drug: Resatorvid
- Resatorvid 2.4 mg/kg/day (Experimental)
  Interventions: Drug: Resatorvid
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Resatorvid — Resatorvid 1.2 mg/kg, injection, subcutaneously for thirty minutes; then resatorvid 0.05 mg/kg/h (1.2 mg/kg/day), injection, subcutaneously over 96 hours.
  Other Names: TAK-242
  Arms: Resatorvid 1.2 mg/kg/day
Drug: Resatorvid — Resatorvid 1.2 mg/kg, injection, subcutaneously for thirty minutes; then resatorvid 0.1 mg/kg/h (2.4 mg/kg/day), injection, subcutaneously over 96 hours.
  Other Names: TAK-242
  Arms: Resatorvid 2.4 mg/kg/day
Drug: Placebo — Resatorvid placebo-matching injection, subcutaneously for thirty minutes; then resatorvid placebo-matching injection, subcutaneously over 96 hours.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the optimal dose of Resatorvid for reducing 28-day all-cause mortality in subjects with severe sepsis.

DETAILED DESCRIPTION:
Severe sepsis, defined as sepsis associated with acute organ dysfunction, remains a serious medical problem worldwide. In the United States alone, approximately 750,000 cases of severe sepsis occur each year, with the mortality rate ranging between 30% and 50% for severe sepsis patients with concomitant organ dysfunction. As the population ages, these numbers are expected to increase. The pathophysiology of severe sepsis is thought to involve the activation of a variety of inflammatory and procoagulant host responses to infection, which if unchecked, can lead to diffuse endovascular injury, multi-organ dysfunction, and ultimately death.

The host response to infection with microorganism and microorganism-derived molecules is characterized by the synthesis and release of pro-inflammatory cytokines such as tumor necrosis factor-alpha (TNF-α) and interleukins 1, 6 and 8 (IL-1, IL-6, and IL-8), by inflammatory cells, and by other markers of inflammation such as C-reactive protein. Inflammatory cells, such as macrophages, release these cytokines by signals transmitted from the surface of these cells after binding of pathogen-associated molecules to cell surface pattern recognition receptors known as toll-like receptors.

TAK-242 (resatorvid) is a small molecule suppressor of pathogen-induced release of inflammatory cytokines and acts by inhibiting TLR-4 mediated signaling. Because of its inhibitory effect on suppressing cytokine levels, resatorvid is being developed as a treatment for severe sepsis.

The study was ended after the DSMB determined there was insufficient cytokine suppression in the 150-subject analysis within Stage 1 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Has clinical evidence of infection defined as the presence of a known or probable source of infection requiring the initiation of parenteral antimicrobial therapy.
* Must meet at least 3 of the following 4 criteria for SIRS:

  * A core temperature greater than 38°C or less than 36°C.
  * A heart rate greater than 90 beats per minute.
  * A respiratory rate greater than 20 breaths/min or partial pressure of carbon dioxide in arterial blood less than 32 mm Hg or mechanical ventilation for an acute process.
  * A total white blood cell absolute count greater than 12,000 cells/mm3 or less than 4,000 cells/mm3, or a white blood cell differential count that showed greater than 10% immature (band) forms.
* Must have sepsis with shock and/or respiratory failure.

Exclusion Criteria

* If female, the subject is pregnant, nursing and the milk is intended to be ingested by the infant, or the participant plans to become pregnant, or nurse and the milk is intended to be ingested by the infant.
* Is receiving immunosuppressive therapy such as cyclosporine, azathioprine, or cancer-related chemotherapy.
* Has a granulocyte count of less than 1000/mm3 except if the decreased count was believed to be due to sepsis.
* Has documented or suspected acute myocardial infarction within the last 6 weeks prior to Pretreatment Period.
* Has a documented history of moderate to severe chronic heart failure as defined by New York Heart Association Functional Classification III or IV.
* Is known to be positive for human immunodeficiency virus with known CD4 count less than or equal to 50/mm3 or had known end-stage processes.
* Has a known history of glucose-6-phosphate dehydrogenase deficiency.
* Has a methemoglobin level greater than 5% at Pretreatment Period or had a known history of methemoglobinemia.
* Is moribund and death was considered imminent.
* Is classified as "Do Not Resuscitate", or "Do Not Treat", or the participant's family has not committed to aggressive management of the participant's condition.
* Is not expected to survive for 28 days and was not likely be given life support due to a pre-existing, uncorrectable medical condition.
* Has a known esophageal varices, chronic jaundice, cirrhosis, or chronic ascites.
* Is in a chronic vegetative state or has a similar long-term neurological condition.
* Has known portal hypertension or Child-Pugh hepatic impairment class C.
* Has acute third degree burns involving more than 30% of body surface within 120 hours prior to Pretreatment Period.
* Has known hypersensitivity to sulfonamides.
* Has known hypersensitivity to components of resatorvid.
* Has participated in any other investigational study (drug or device) and/or taken any investigational drug within 30 days or 5 half-lives of the drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2005-09; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
28-day All-cause Mortality. | Day 28

SECONDARY OUTCOMES:
Change from Baseline in Organ Failure Assessment | Day 28
Mean Systemic Inflammatory Response | Day 28
Mean Vasopressor-free days | Day 28
Mean Ventilator-free days | Day 28
Mean Intensive Care Unit free days | Day 28
Mean Discharge Status. | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science, Study Director — Takeda
Locations (144):
- United States (49):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Escondido, California
  - Los Angeles, California
  - Orange, California
  - Poway, California
  - San Diego, California
  - Colorado Springs, Colorado
  - New Haven, Connecticut
  - Newark, Delaware
  - Atlantis, Florida
  - Bay Pines, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Sarasota, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - Peoria, Illinois
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Louisville, Kentucky
  - Shreveport, Louisiana
  - Portland, Maine
  - Baltimore, Maryland
  - Springfield, Massachusetts
  - Kalamazoo, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Butte, Montana
  - Englewood, New Jersey
  - Buffalo, New York
  - New York, New York
  - Rochester, New York
  - Greensboro, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Greenville, South Carolina
  - Nashville, Tennessee
  - Fort Worth, Texas
  - Galveston, Texas
  - Houston, Texas
  - Lubbock, Texas
  - Bellevue, Washington
- Australia (3):
  - Adelaide
  - Fremantle
  - Heidelberg
- Austria (2):
  - Linz
  - Vienna
- Belgium (8):
  - Aalst
  - Antwerp
  - Brussels
  - Genk
  - Ghent
  - Liège
  - Ottignies
  - Yvoir
- Canada (6):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - London, Ontario
- Czechia (6):
  - Brno
  - Havlíčkův Brod
  - Hradec Králové
  - Opava
  - Pilsen
  - Prague
- Finland (9):
  - Helsinki
  - Joensuu
  - Kokkola
  - Kuopio
  - Lappeenranta
  - Oulu
  - Seinäjoki
  - Tampere
  - Turku
- Germany (9):
  - Berlin
  - Dresden
  - Erfurt
  - Jena
  - Krefeld
  - Ludwigshafen
  - Mannheim
  - München
  - Wuppertal
- Israel (8):
  - Afula
  - Ashkelon
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Ẕerifin
- Italy (3):
  - Lecco
  - Monza
  - Pavia
- Japan (11):
  - Chiba
  - Fukuoka
  - Hiroshima
  - Hokkaido
  - Kumamoto
  - Kyoto
  - Numakunai
  - Osaka
  - Shizuoka
  - Tokyo
  - Yamaguchi
- Netherlands (7):
  - 's-Hertogenbosch
  - Apeldoorn
  - Groningen
  - Leeuwarden
  - Nijmegen
  - Rotterdam
  - Tilburg
- New Zealand (4):
  - Auckland
  - Christchurch
  - Hastings
  - Tauranga
- San Juan, Puerto Rico
- Spain (5):
  - Barcelona
  - Getafe
  - Madrid
  - Valladolid
  - Vitoria-Gasteiz
- Sweden (8):
  - Gävle
  - Gothenburg
  - Karlstad
  - Kristianstad
  - Linköping
  - Lund
  - Stockholm
  - Uppsala
- United Kingdom (5):
  - Brighton
  - Glasgow
  - Leeds
  - Livingston
  - London

REFERENCES:
- [Result] Rice TW, Wheeler AP, Bernard GR, Vincent JL, Angus DC, Aikawa N, Demeyer I, Sainati S, Amlot N, Cao C, Ii M, Matsuda H, Mouri K, Cohen J. A randomized, double-blind, placebo-controlled trial of TAK-242 for the treatment of severe sepsis. Crit Care Med. 2010 Aug;38(8):1685-94. doi: 10.1097/CCM.0b013e3181e7c5c9. PMID 20562702